CLINICAL TRIAL: NCT00624676
Title: Randomized Study Comparing the Efficacy and Tolerance of a Lipophilic Hydroxy Acid Derivative of Salicylic Acid and 5% Benzoyl Peroxide in the Treatment of Facial Acne Vulgaris
Brief Title: Efficacy and Tolerance of a Derivative of Salicylic Acid and 5% Benzoyl Peroxide in Facial Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Principal Investigator, Robert BISSONNETTE, President and Dermatologist, Cosmetique Active International
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LRP05021
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Acne Vulgaris
Keywords: Acne; lipophilic hydroxy acid; benzoyl peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — capryloyl salicylic acid; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): LHA formulation
  Interventions: Drug: Lipo Hydroxy Acid
- B (Active Comparator): 5% benzoyl peroxide
  Interventions: Drug: 5% benzoyl peroxide gel

INTERVENTIONS:
Drug: Lipo Hydroxy Acid — Twice a day
  Other Names: Effaclar AI; 2-hydroxy 5-octanoyl benzoic acid; LHA; C8-LHA; capryloyl salicylic acid
  Arms: A
Drug: 5% benzoyl peroxide gel — Once a day
  Other Names: PanOxyl 5
  Arms: B

SUMMARY:
Acne vulgaris is a frequent inflammatory skin condition involving the pilosebaceous unit and affecting more than 80% of teenagers. Mild to moderate acne vulgaris is usually treated with topical agents such as benzoyl peroxide, retinoids and antibiotics. These treatments can be associated with local tolerance problems and/or antibiotic resistance. Salicylic acid has been shown to be an effective treatment for acne. LHA is a lipophilic hydroxy acid derivative of salicylic acid that has comedolytic and antibacterial properties.

The objective of this trial was to compare the efficacy and tolerance of a cream formulation containing 0.3% LHA (LHA formulation) to a 5% benzoyl peroxide gel.

DETAILED DESCRIPTION:
This was a randomized clinical trial performed at two centers (Montreal and Laval, Quebec, Canada) under the direction of the same principal investigator. Eighty (80) subjects were enrolled in the study. Subjects were asked to report to the clinic for four visits (D0, D28, D56, D87). The LHA formulation was applied twice a day (morning and evening) and benzoyl peroxide was applied daily (evening) on a clean face for a total of 12 weeks.

Efficacy was evaluated at day 28, 56 and 87. The number of papules, pustules, opened and closed comedones were counted at each visit by a blinded assessor. The overall efficacy was evaluated with a 4-point scale (no improvement, moderate, good and excellent) by the subject and the blinded assessor. Clinical examination included evaluation of sensitivity of the skin (presence of erythema and desquamation) by the investigator and of pruritus, tingling and burning sensation by subjects on a 4-point scale. Finally, the subject and the skin assessor both evaluated overall tolerance on a 4-point scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Phototype greater than I
* Facial inflammatory acne with 15-50 inflammatory lesions and less than 50 non-inflammatory lesions (excluding the nasal pyramid)
* Did not receive a topical acne treatment in the last 15 days
* Did not receive cyclins or zinc-based treatment in the last month
* Did not take Diane-35 in the last 2 months. Current use of oral contraceptives is acceptable if the subject is on a stable dose for at least six months prior Day 0.
* Did not take oral isotretinoin for the last 12 months
* Did not change their cosmetic habits in the last 15 days (ex: shaving cream)
* Agree to participate to the entire study

Exclusion Criteria:

* Less than 18 years old
* Phototype I
* With less than 15 or more than 50 inflammatory lesions on the face (excluding the nasal pyramid)
* With more than 50 non-inflammatory lesions on the face (excluding the nasal pyramid)
* Have taken 1) A topical acne treatment in the last 15 days, or 2) Cyclins or zinc-based treatment in the last month or 3) Oral isotretinoin in the last 12 months
* Woman: 1) Taking Diane-35, or 2) Taking an oral contraceptive for less than 6 months or 3) That are pregnant or 4) That are nursing or 5) Not using any efficient contraception method (if necessary)
* With a history of allergic reaction or hypersensitivity to one of the constituents of the study product
* With peroxide sensitivity
* With history of photosensitivity
* With history of major medical or psychiatric condition or surgical interventions that, in the opinion of the investigator, might put the subject at risk
* With an acute or chronic disease that could interfere with study results
* Susceptible to take a corticosteroid treatment during the study except inhaled or topic when needed to treat a condition outside the face
* With a dermatologic condition on the face other than acne that might put the subject at risk or interfere with study evaluations
* Using another cosmetic product than the one received for this study. Sunscreens are allowed occasionally.
* Subject who must have extensive sun or ultra-violet exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Reduction in inflammatory lesions | Days 28, 56 and 87

SECONDARY OUTCOMES:
Reduction in non-inflammatory lesions | Days 28, 56 and 87
Overall efficacy | Days 28, 56 and 87
Overall tolerance | Days 28, 56 and 87
Evaluation of pruritus, burning and tingling by the subject | Days 28, 56 and 87
Evaluation of erythema and desquamation by the blind assessor | Days 28, 56 and 87

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research
Locations (2):
- Canada (2):
  - Innovaderm Research, Laval, Quebec
  - Innovaderm Research, Montreal, Quebec